CLINICAL TRIAL: NCT05101980
Title: Predictors of Atrial Fibrillation Recurrence After Ablation Using PENTARAY Catheter
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maria Hamdy Bassit, Maria Bassit, Assiut University
Other Study IDs: PENTARAY catheter
Record Dates: First submitted 2021-10-20; First posted 2021-11-01 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Atrial Fibrillation Ablation Using PENTARAY Catheter

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
CARTO represent a new way of 3D electroanaromic mapping for AF which has improved safety and success rate of AF ablation compared with other conventional methods of AF ablation as it provide accurate visualization of atrial anatomy and identification of atrial substrate properties for catheter ablation of atrial arrythmias which ensure good ablation with decreased incidence of recurrence of AF.

ELIGIBILITY:
Inclusion Criteria:

* Patient with paroxismal AF who are eligible for AF ablation
* Patient resistant to medical treatment

Exclusion Criteria:

* Patient with other types of arrythmias
* Patient with prothetic valves
* Patient with valvular AF

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with paroxismal AF who are eligible for AF ablation
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Maintenance of sinus rhythm after successful ablation of atrial fibrillation | 6 months after AF ablation